CLINICAL TRIAL: NCT02023775
Title: Non Interventional Study on Pulmonary Valve Replacement by Thranscatheter Pulmonary Valve Melody™
Acronym: Melody™FR
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Melody™ France
Record Dates: First submitted 2013-04-29; First posted 2013-12-30 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2020-09

CONDITIONS: Right Ventricular Congenital Cardiopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients implanted with Medtronic Melody valve: All patients that received a valve implantation were included in the registry.
  Interventions: Device: Melody valve implantation

INTERVENTIONS:
Device: Melody valve implantation

SUMMARY:
Prospective, longitudinal, open-label, multicentre, observational, non-comparative national study using an exhaustive registry of implantations over a given period.

This study is requested by French Health Authorities for reimbursement renewal, to maintain reimbursement for pulmonary valvular replacement by bioprothesis in approved indication in France.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, open-label, multicentre, observational, non-comparative national study using an exhaustive registry of implantations over a given period in France. The study is requested by French Health Authorities in 2010 for reimbursement renewal, to maintain reimbursement for pulmonary valvular replacement by bioprothesis in approved indication in France. The study was closed in 2013.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring pulmonary valvular replacement for correction of right ventricular ejection path malfunction (stenosis and/or pulmonary regurgitation).

Exclusion Criteria:

* Patient or legal representative refusal to data collection or processing
* Patient unable to guarantee follow-up data collection, in particular for patients living abroad

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients receiving a valve implantation, without exception (exhaustive population)
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2010-01-31 (Actual); Primary Completion 2013-01-24 (Actual); Study Completion 2013-10-20 (Actual)

PRIMARY OUTCOMES:
absence of re-intervention on the pulmonary valve | 12 months
  to evaluate the efficacy of the MELODY valve, defined as the absence of re-intervention on the pulmonary valvee

SECONDARY OUTCOMES:
rate re-intervention on the valve | 60 months
  To document the rate re-intervention on the valve during a 60 months follow-up after its implantation
time period before re-intervention on the valve | 60 months
  To document the time period before re-intervention on the valve (longevity of the prosthesis), the reasons for re-intervention (stent fracture, leak, stenosis) and the rate of durability (% of implanted valves with malfunction requiring a re-intervention)
patient characteristics | 60 months
  To compare the patient characteristics to the indications of the bioprosthesis
Description and time of onset of open surgery after implantation | 60 months
  Description and time of onset of open surgery after implantation on first implanted patients versus device replacement
failures of the implantation procedure | 60 months
  To document the failures of the implantation procedure
survival rate at 12, 36, 48 and 60 months | 60 months
  To document the survival rate at 12, 36, 48 and 60 months
frequency of antiplatelet treatment during and after implant | 60 months
  To describe the frequency of antiplatelet treatment during and after implant
patients' characteristics to indications of the MELODY™ bioprosthesis | 60 months
  To compare patients' characteristics to indications of the MELODY™ bioprosthesis
time period before the resumption of professional, university or scholastic activity | 60 months
  To document the time period before the resumption of professional, university or scholastic activity

CONTACTS AND LOCATIONS:
Overall Officials: Sophie MALEKZADEH-MILANI, MD, Principal Investigator — Hôpital des enfants Malades - Necker, 149 rue de Sèvres, 75015 Paris, France
Locations (10):
- France (10):
  - Hôpital Louis Pradel, Bron
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Centre chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Hôpital Cardiologique, Lille
  - Hôpital de La Timone Enfants, Marseille
  - Hôpital Laënnec, Nantes
  - Hôpital des enfants Malades Necker, Paris
  - Hôpital Cardiologique du Haut-Lévêque, Pessac
  - Hôpital des enfants Purpan, Toulouse
  - Clinique Pasteur, Toulouse